CLINICAL TRIAL: NCT03943576
Title: Adipose-Derived Stem Cells (ADSCs) Injections for Knee Osteoarthritis
Brief Title: Allogeneic Adipose Tissue-Derived Mesenchymal Stem Cells (GXCPC1) for Knee Osteoarthritis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gwo Xi Stem Cell Applied Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GXCPC1
Record Dates: First submitted 2019-01-23; First posted 2019-05-09 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GXCPC1 (Experimental): GXCPC1 contains 6.7×10^6 or 4×10^7 allogeneic adipose-derived stem cells (ADSCs) in 3 mL
  Interventions: Drug: GXCPC1
- hyaluronic acid (Active Comparator): Hya Joint Plus synovial fluid supplement 3mL
  Interventions: Device: HA

INTERVENTIONS:
Drug: GXCPC1 — The dose regimen is one single intra-articular injection of GXCPC1 containing 6.7×10^6 or 4×10^7 ADSCs in 3 mL saline. (allogeneic injection)
  Arms: GXCPC1
Device: HA — Hya Joint Plus synovial fluid supplement 3mL
  Arms: hyaluronic acid

SUMMARY:
The aim of the investigators study was to investigate the safety and efficacy of allogeneic ADSCs for the clinical treatment of knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Aged 40 to 80 years old (inclusive)
3. Kellgren-Lawrence grading II-IV, as determined by American College ofRheumatology (ACR) criteria for osteoarthritis of the knee
4. Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain score of 7 ~ 17 (inclusive) in the target knee despite use of NSAID
5. Contraindicated to long term systemic NSAID (e.g. suffer from severe gastrointestinal side effects upon systemic NSAID administration, or due to underlying increased gastrointestinal, cardiovascular, or renal risk) and not able to receive or wish to delay knee arthroplasty

Exclusion Criteria:

1. With previous surgery of articular fracture, ligament reconstruction, meniscal reconstruction, and knee arthroplasty on the target knee joint
2. With previous intra-articular intervention (e.g. steroid, anesthetics, hyaluronate, arthroscopic surgery) on the target knee joint 12 weeks prior to screening
3. Administered or required systemic or local on the target knee joint immunosuppressive agent, anti-inflammatory drug, steroid, analgesics, opioid, or duloxetine for OA knee except for acetaminophen and NSAID within 1 week prior to screening
4. With joint diseases other than knee osteoarthritis considered by investigator not eligible to enter the study
5. Unable to receive MRI examination, including allergic to the contrast medium for MRI used in the study, with known history of claustrophobia, having any existing metallic intraocular foreign body or active/inactive implanted medical devices, such as cardiac pacemaker, cochlear, intracranial vascular clips or neurostimulator
6. Active or suspected infection of the target knee joint
7. History of human immunodeficiency virus (HIV) infection
8. History of malignancy within 2 years prior to screening
9. With body mass index (BMI) greater or equal to 35 kg/m2
10. Known hypersensitivity to any component of the investigational product or the active control
11. Participated other investigational study within 4 weeks prior to screening
12. With ongoing or within the past 2 years serious medical conditions (e.g. concomitant illness) such as cardiovascular (e.g. New York Heart Association grade III or IV), hepatic (e.g. Child-Pugh Class C), psychiatric condition (e.g. alcoholism, drug abuse), medical history, physical findings, or laboratory abnormality that in the investigators' opinion could interfere with the results of the trial or adversely affect the safety of the subject
13. Female subject with childbearing potential who is lactating or has positive serum or urine pregnancy test at Screening
14. Subject with childbearing potential refuses to use highly effective contraceptives from signing informed consent until Final/Early Termination Visit. At least two forms of birth control must be adopted and one of which must be a barrier method. Acceptable forms include:

    * Established use of oral, injected or implanted hormonal methods of contraception
    * Placement of an intrauterine device (IUD) or intrauterine system (IUS)
    * Barrier methods of contraception: condom, or occlusive cap (diaphragmor cervical/vault caps)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2022-04-27 (Actual); Study Completion 2023-03-22 (Actual)

PRIMARY OUTCOMES:
WOMAC pain score | week 24
  Change from baseline in WOMAC pain score at Week 24

SECONDARY OUTCOMES:
MRI | week 0, 24, 48
  Change from baseline to post-treatment visits on the target knee in MRI examination results
Visual Analogue Scale (VAS) | week 0, 1, 4, 12, 24
  Changes from baseline to post-treatment visits on the target knee in Visual Analogue Scale (VAS) for pain
12-item Short Form (SF-12) | week 0, 1, 4, 12, 24
  Change from baseline to post-treatment visits in total score of 12-item Short Form (SF-12) health survey questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-FONG Chen, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- GWOXI Stem Cell Applied Technology Co., Ltd., Hsinchu, Taiwan

REFERENCES:
- [Derived] Chen CF, Chen YC, Fu YS, Tsai SW, Wu PK, Chen CM, Chen WM, Wu HH, Lee CH, Chang CL, Lin PC, Kao YC, Chen CH, Chuang MH. Safety and Tolerability of Intra-Articular Injection of Adipose-Derived Mesenchymal Stem Cells GXCPC1 in 11 Subjects With Knee Osteoarthritis: A Nonrandomized Pilot Study Without a Control Arm. Cell Transplant. 2024 Jan-Dec;33:9636897231221882. doi: 10.1177/09636897231221882. PMID 38205679